CLINICAL TRIAL: NCT01009476
Title: Non-interventional Study on Long-term Application of Galantamine and Nootropics in Patients With Alzheimer's Disease
Brief Title: Long-term Use of Galantamine Versus Nootropics (Memory Enhancing Drugs) in Patients With Alzheimer's Dementia Under Conditions of Daily Routine
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor
Other Study IDs: CR011689
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Dementia; Alzheimer Disease; Dementia, Vascular
Keywords: Dementia; Galantamine; Cholinesterase inhibitors; Nootropic agents; Alzheimer; Vascular dementia; Cognitive symptoms; Behavioural symptoms; Care giving times
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular; Neurobehavioral Manifestations; Behavioral Symptoms | interventions — Galantamine; Nootropic Agents; Ginkgo Extract; Nicergoline; Piracetam

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 001
  Interventions: Drug: Galantamine
- 002
  Interventions: Drug: Nootropics (ginkgo biloba, nicergoline, piracetam, or others)

INTERVENTIONS:
Drug: Galantamine — Therapeutic measures were not predefined in the protocol but remained at the discretion of the treating physician. The treatment regimen of galantamine (8 mg,16 mg, 24 mg retard capsule) was to be in accordance with the recommendations given in the summary of product characteristics.
  Groups: 001
Drug: Nootropics (ginkgo biloba, nicergoline, piracetam, or others) — Therapeutic measures were not predefined in the protocol but remained at the discretion of the treating physician. The treatment regimen of nootropics was to be in accordance with the recommendations given in the relevant summary of product characteristics.
  Groups: 002

SUMMARY:
The main objective of this non-interventional study was to document the long-term application of galantamine and nootropics (memory enhancing drugs) over a period of 1 year under conditions of daily routine. There were no predefined specifications of diagnostic and therapeutic measures. The decision for treatment with either galantamine or a nootropic had to be made by the treating physician prior to the start of documentation. The following measures were to be documented: safety, tolerability, dementia-associated symptoms (unstable walking, vertigo, awakening at night, shouting/screaming at night, perambulating at night, aggressiveness, agitation, apathy/social retreat, delusions, hallucinations, behavior that poses a risk to self or others, and daytime tiredness), frequency of admissions to nursing homes or nursing services, global functional level, caregiver's burden, and time spent on caregiving. Furthermore, this study aimed to gather knowledge on the differentiated use of the two treatment strategies considering the specific diagnosis of dementia (e.g. Alzheimer's disease only or mixed dementia, i.e. Alzheimer's disease and cerebrovascular disease) and risk profiles.

DETAILED DESCRIPTION:
The aim of this observational, non-interventional study was to observe and document for a 1-year period, the long-term use of galantamine and nootropics (memory enhancing drugs) over a 1 year period under conditions of daily routine in a typical patient population of patients with mild or moderate Alzheimer's dementia or with mixed dementia, i.e. Alzheimer's and cerebrovascular disease. The design of this prospective study was non-interventional and thus, there were no predefined specifications of diagnostic and therapeutic measures. The decision for treatment with either galantamine or a nootropic agent had to be made by the treating physician prior to the start of documentation. Patients were observed over a period of 12 months or until end of documentation (visit 1 = baseline; visit 2, 3 and 4 after approximately 2, 6 and 9 months, respectively; visit 5 after approximately 12 months or final visit at end of documentation). The following measures were to be documented: safety by documenting adverse and serious adverse events together with severity, outcome and causality to the treatment; tolerability; vital functions; Global Deterioration Scale (GDS) staging system assessing global functioning; Mini-Mental State Examination assessing cognitive functions; dementia-associated behavioural symptoms (unstable walking, vertigo, awakening at night, shouting/screaming at night, perambulating at night, aggressiveness, agitation, apathy/social retreat, delusions, hallucinations, behavior that poses a risk to self or others, and daytime tiredness); frequency of admissions to nursing homes or nursing services; caregiver's burden and time spent on caregiving (based on daily and weekly caregiving tasks); final evaluation of the therapy with galantamine or nootropics through the treating physician. Furthermore, this study aimed to gather knowledge on the differentiated use of the two treatment strategies considering the specific diagnosis of dementia (e.g. Alzheimer's disease only or mixed dementia, i.e. Alzheimer's disease and cerebrovascular disease) and risk profiles. Therapeutic measures were not predefined in the protocol but remained at the discretion of the treating physician. Therapy decisions were to be based on medical needs. The treatment regimen of galantamine (8 mg,16 mg, 24 mg retard capsule) or nootropic agents (e.g. ginkgo biloba, dihydroergotoxine, nicergoline, piracetam, or others) was to be in accordance with the recommendations given in the summary of product characteristics (SmPC).

ELIGIBILITY:
Inclusion Criteria:

* Patients were selected for documentation after the decision of treatment (galantamine or nootropic) had been made by the treating physician. Patients documented in this study were required to meet the following selection criteria: Diagnosis of probable mild or moderate dementia: Alzheimer type or mixed dementia (Alzheimer's and cerebrovascular disease)
* Mini-Mental-State Examination score = 24 at baseline (Visit 1), if possible
* Monotherapy with either galantamine or nootropic (the decision for treatment with either galantamine or a nootropic had to be made by the treating physician prior to the start of documentation)
* Patient had a caregiver to whom personal contact was possible at least 3 times per week

Exclusion Criteria:

* Patients were not eligible if they had received anti-dementive treatment with acetylcholinesterase inhibitors, memantine, or the same nootropic used during the observational period within the last 12 weeks prior to baseline

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mild or moderate Alzheimer dementia with or without cerebrovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 1134 (Actual)
Dates: Start 2006-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
documentation of the long-term use of galantamine and nootropics over a 1 year period under conditions of daily routine in patients with Alzheimer's disease (with or without vascular pathology) | approx. 12 months or until end of observation ( visit 1 = baseline; visit 2, 3 and 4 after approximately 2, 6 and 9 months, respectively; visit 5 after approximately 12 months or final visit at end of documentation)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag G.m.b.H. Clinical Trial, Study Director — Janssen-Cilag G.m.b.H